CLINICAL TRIAL: NCT03239028
Title: Dietary Quality During Adolescence is Associated With Mother's Dietary Quality During Pregnancy: 15 Years Follow up From a Large National Birth Cohort
Brief Title: Dietary Quality During Adolescence is Associated With Mother's Dietary Quality During Pregnancy
Status: Completed | Type: Observational
Sponsor: Centre for Fetal Programming, Denmark (Other)
Collaborators: Statens Serum Institut (Other); University of Iceland (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-04 M-C Association
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Eating Behavior
Keywords: diet quality; pregnancy; adolescence; longitudinal study; food frequency questionnaire
MeSH Terms: conditions — Feeding Behavior | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish National Birth Cohort
  Interventions: Behavioral: Observational

INTERVENTIONS:
Behavioral: Observational

SUMMARY:
We will examine the association between diet quality in offspring at age 14 years and maternal diet quality during pregnancy in the Danish National Birth Cohort

DETAILED DESCRIPTION:
Background: Dietary exposures in fetal life may have long lasting impact on the individual's susceptibility for several non-communicable diseases. Although offspring's own dietary habits become increasingly independent from parental influence other external factors are likely to exist. Further insights are needed to interpret and separate potential influence from exposures in pregnancy from later dietary habits on later disease risk.

Objectives: We will examine the association between diet quality in offspring at age 14 years and maternal diet quality during pregnancy in the Danish National Birth Cohort (DNBC).

Design: A total of 19620 DNBC offspring-mother pairs will be matched by offspring dietary intake assessed at age ~14 years with a 150-item food frequency questionnaire (FFQ) and dietary intake assessed with a 300-item FFQ during mid-pregnancy (1996-2003). A Healthy Eating Index (HEI) will be developed as an indicator for diet quality based on current Danish Food-Based Dietary Guidelines including 8 components; fruit and vegetables, fish, dietary fibers, red meat, saturated fatty acids, sodium, sugar-sweetened beverages, and added sugar.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the Danish National Birth Cohort

Exclusion Criteria:

* If mother did not complete a food frequency questionnaire during pregnancy

Ages: 14 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Around 95,000 children born during 1996-2003 in Denmark were recruited for The Danish National Birth Cohort
Sampling Method: Non-Probability Sample
Enrollment: 19620 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Diet quality | Reported intake during one year
  Healthy Eating Index depicting diet quality

CONTACTS AND LOCATIONS:
Overall Officials: Sjurdur F Olsen, PhD, Study Director — Statens Serum Institut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Olsen J, Melbye M, Olsen SF, Sorensen TI, Aaby P, Andersen AM, Taxbol D, Hansen KD, Juhl M, Schow TB, Sorensen HT, Andresen J, Mortensen EL, Olesen AW, Sondergaard C. The Danish National Birth Cohort--its background, structure and aim. Scand J Public Health. 2001 Dec;29(4):300-7. doi: 10.1177/14034948010290040201. PMID 11775787
- [Result] Olsen SF, Mikkelsen TB, Knudsen VK, Orozova-Bekkevold I, Halldorsson TI, Strom M, Osterdal ML. Data collected on maternal dietary exposures in the Danish National Birth Cohort. Paediatr Perinat Epidemiol. 2007 Jan;21(1):76-86. doi: 10.1111/j.1365-3016.2007.00777.x. PMID 17239183
- See also: Link to web-page of Centre for Fetal Programming — http://www.cfp-research.com/